CLINICAL TRIAL: NCT06886243
Title: Effect of Menstrual Cycle on Postoperative Sensitivity and Rebound Pain in Posterior Composite Restorations: A Double-Blind Split-Mouth Clinical Study
Brief Title: Menstrual Cycle Effects on Postoperative Sensitivity and Rebound Pain in Composite Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Adem GOK, DDs, PhD, Assistant Professor, Firat University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FIRAT-DENTISTRY ADEMGOK-001; 1919B012224148 (Other Grant/Funding Number: TUBİTAK)
Record Dates: First submitted 2025-03-09; First posted 2025-03-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Sensitivity; Rebound Pain; Menstrual Cycle; Composite Restorations

STUDY DESIGN:
Intervention Model Description: This study is designed as a double-blind, split-mouth, randomized clinical trial. Each participant undergoes two direct posterior composite restorations in different menstrual cycle phases.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Both the operator performing the restorations and the researcher assessing postoperative sensitivity and rebound pain were blinded to the menstrual cycle phases of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Menstrual Phase Group (MPG) (Experimental): Arm 1: Menstrual Phase Group (MPG) Arm Type: Experimental Arm Name: Menstrual Phase Group (MPG) Description: Participants receive a direct posterior composite restoration during the menstrual phase of their cycle. Postoperative sensitivity (POS) and rebound pain (RP) are assessed at multiple time points.
  Interventions: Procedure: Direct Posterior Composite Restoration
- Ovulatory Phase Group (OPG) (Experimental): Arm 2: Ovulatory Phase Group (OPG) Arm Type: Experimental Arm Name: Ovulatory Phase Group (OPG) Description: Participants receive a direct posterior composite restoration during the ovulatory phase of their cycle. POS and RP are assessed at multiple time points.
  Interventions: Procedure: Direct Posterior Composite Restoration

INTERVENTIONS:
Procedure: Direct Posterior Composite Restoration — Description: Composite restorations performed using Clearfil Majesty Posterior (Kuraray, Japan) and Clearfil Universal Bond Quick (Kuraray, Japan) in self-etch mode.
  Inferior alveolar nerve block (IANB) administered with articaine hydrochloride with epinephrine (1:100,000) (Maxicaine).

SUMMARY:
This study aims to evaluate how different phases of the menstrual cycle affect pain after dental treatments. Specifically, it investigates two types of pain:

Postoperative sensitivity (pain felt after the filling procedure), and Rebound pain (pain that begins after the numbness from anesthesia wears off). The study was conducted with 35 women who received two dental fillings at different times in their cycle: once during the menstrual phase and once during the ovulatory phase.

A local anesthetic (inferior alveolar nerve block) was used before treatment, and pain was measured using a 0-10 visual scale at several time points after the procedure.

The goal of the study is to understand whether hormonal changes during the menstrual cycle can affect pain levels after dental work. This information could help dentists improve pain management strategies for women and personalize treatment timing.

DETAILED DESCRIPTION:
This clinical trial investigates the effect of menstrual cycle phases on postoperative pain perception following direct posterior composite restorations. It addresses the hypothesis that hormonal fluctuations during the menstrual cycle may alter pain thresholds and nociceptive processing, potentially influencing the intensity and timing of postoperative dental pain.

Estrogen and progesterone, the primary hormones involved in the menstrual cycle, have been shown to modulate pain through their effects on the central and peripheral nervous systems, inflammatory mediators, and endogenous opioid pathways. Despite extensive research on hormonal influences in systemic pain, their specific effects on dental pain-particularly postoperative sensitivity and rebound pain-remain understudied.

The study employed a double-blind, split-mouth, randomized clinical design to minimize inter-subject variability and strengthen internal validity. A total of 35 female participants with regular menstrual cycles underwent two posterior Class II composite restorations, one during the menstrual phase (MPG) and one during the ovulatory phase (OPG). Menstrual phases were confirmed using self-reported cycle calendars and mobile tracking applications.

All restorative procedures were standardized and performed under local anesthesia. Composite restorations were completed using Clearfil Majesty Posterior and Clearfil Universal Bond Quick (self-etch mode). An inferior alveolar nerve block (IANB) was administered using articaine hydrochloride with epinephrine (1:100,000).

Pain was assessed using the Visual Analog Scale (VAS, 0-10) at predefined time points to evaluate two types of postoperative discomfort:

Postoperative Sensitivity (POS): assessed on Day 1, Day 2, and Day 3 following the procedure.

Rebound Pain (RP): assessed at Hour 4, Hour 8, and Hour 12 after the resolution of anesthesia.

Statistical analyses were performed using Cochran's Q test and McNemar's test for within-subject comparisons, and Chi-Square or Fisher's Exact Test for between-group differences. Bonferroni correction was applied for multiple comparisons to control type I error, with p < 0.05 considered statistically significant.

This study provides new insights into the chronobiological factors affecting dental pain and contributes to the evidence base for individualized pain management in female dental patients. The findings may support more personalized scheduling of restorative procedures and better prediction of analgesic needs based on menstrual cycle phases.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18-45 years
* Regular naturally occurring menstrual cycles (26-32 days)
* No use of hormonal contraceptives
* Good general health
* Vital posterior molar teeth requiring direct composite restorations
* Good oral hygiene and periodontal health

Exclusion Criteria:

* Irregular menstrual cycles or known hormonal disorders
* Presence of dentin hypersensitivity in the affected tooth
* Regular use of psychiatric or other medications
* History of bruxism, temporomandibular disorders (TMD), or chronic pain syndromes Pregnancy or lactation
* Use of analgesics, oral contraceptives, or anti-inflammatory drugs within 48 hours before treatment
* Severe periodontal disease, dental pain, or need for endodontic treatment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is limited based on biological sex due to menstrual cycle-related variables
Enrollment: 35 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Sensitivity (POS) Score Measured Using Visual Analog Scale (VAS) | Day 1, Day 2, and Day 3 after restoration
  Postoperative sensitivity (POS) is assessed using the Visual Analog Scale (VAS, 0-10).
  A score of 0 represents no pain/sensitivity, while 10 represents unbearable pain/sensitivity.
  Clinically significant postoperative sensitivity is defined as VAS ≥4. Measurements are recorded at 24, 48, and 72 hours after the restoration. Description: Postoperative sensitivity (POS) will be evaluated using the Visual Analog Scale (VAS, 0-10), where 0 represents no pain/sensitivity and 10 represents unbearable pain/sensitivity. Sensitivity will be recorded at 24, 48, and 72 hours postoperatively. A VAS score ≥4 will be considered clinically significant.

SECONDARY OUTCOMES:
Rebound Pain (RP) Score Measured Using Visual Analog Scale (VAS) | Hour 4, Hour 8, and Hour 12 after anesthesia resolution.
  Rebound pain (RP) is assessed using the Visual Analog Scale (VAS, 0-10) at predefined intervals after the anesthetic effect resolves.
  A score of 0 represents no pain, while 10 represents the worst pain experienced.
  Clinically significant rebound pain is defined as VAS ≥4. Measurements are recorded at 4, 8, and 12 hours postoperatively after anesthesia resolution.

CONTACTS AND LOCATIONS:
Locations (1):
- Firat University Faculty of Dentistry, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share individual participant data.

REFERENCES:
- [Background] Eshghpour M, Rezaei NM, Nejat A. Effect of menstrual cycle on frequency of alveolar osteitis in women undergoing surgical removal of mandibular third molar: a single-blind randomized clinical trial. J Oral Maxillofac Surg. 2013 Sep;71(9):1484-9. doi: 10.1016/j.joms.2013.05.004. Epub 2013 Jul 15. PMID 23866782

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT06886243/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT06886243/ICF_001.pdf